CLINICAL TRIAL: NCT04474288
Title: SARS-CoV-2 Specific Immune Responses in Hospitalized Persons Under Investigation (PUIs) With Negative Nasopharyngeal PCR Swabs - The COVID-19 PUI Reality Check (CPRC) Study
Brief Title: The COVID-19 PUI Reality Check (CPRC) Study
Acronym: CPRC
Status: Completed | Type: Observational
Sponsor: Bassett Healthcare (Other)
Collaborators: Bioreference, Inc (Unknown)
Responsible Party: Principal Investigator, Daniel Freilich, MD, attending physician - hospitalist/infectious disease, Bassett Healthcare
Other Study IDs: 1613182
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Covid19 Immunology
MeSH Terms: interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Biospecimens will be analyzed to assess antibody levels, RNA analysis, and analysis of other immunological markers. Subjects have the option to allow their specimens to be retained for future designated research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Person Under Investigation (PUI): PUI's are subjects who were admitted to the hospital with symptoms suspicious for COVID-19.
  Interventions: Diagnostic Test: SARS-CoV-2 antibody testing
- Asymptomatic Person under Screening (APS): APS's are those patients who do NOT meet the criteria to be a suspect COVID- 19 patient but are being tested because they are being admitted, are required for testing by state mandate, or are having a procedure, etc.
  Interventions: Diagnostic Test: SARS-CoV-2 antibody testing

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 antibody testing — venipuncture for SARS-CoV-2 IgG

SUMMARY:
This study compares SARS-CoV-2 immune responses in high pretest probability swab negative hospitalized PUI patients vs. low pretest probability swab negative hospitalized APS (Asymptomatic Persons being Screened) patients to try to understand the appropriateness and safety of clinical decisions made in these patient populations based on swab results.

DETAILED DESCRIPTION:
This is essentially a two phase blood drawing and immune assays study. Phase 1 will be a single convalescent timing immune retrospective study; phase 2 will include paired samples to increase immune response accuracy in a prospective study. In phase 1, hospitalized PUI and APS patients with negative nasopharyngeal PCR swabs selected by Epic query of Bassett records, will be contacted by telephone (or in person if hospitalized), offered enrollment in the study, and provided informed consent if they're interested. For consented/enrolled patients, routine baseline demographic and clinical data will be obtained by interview (in person or telephone) and/or EMR (Epic) review. These data will be needed to describe baseline characteristics and to assess for predictors of serologic conversion and other immune responses in the two study populations. Up to two to three visits will be required for brief interviews, record review, and blood draws. Phase 1 patients will have visits/blood draws on days 14 and 28 after hospitalization or at 28 days after hospitalization only (-3 days, +60 days) if patients are beyond day 14 at the time of study initiation; phase 2 patients will have visits/blood draws aiming for days 0, 14 (+/- 3 days), and 28 (+/- 3 days) after hospital admission.

Blood will be drawn for SARS-CoV-2 specific immune assays (below). For phase 1 patients, baseline immune assays will not be available as blood is not available for them; thus, for many phase 1 patients, only one of the day 14 and 28 immune assays will be practical. In Phase 2, these procedures will be the same except baseline blood draws will be possible at hospitalization as well. Thus, blood drawing will be at target days 0, 14, and 28 for phase 2 patients. Short interviews at days 14 and 28 will be conducted to assess for new COVID-19 compatible illnesses that may confound immune response results.

Up to 27.5 ml of blood will be required at each timepoint (PAXgene tube 2.5 ml, heparinized tube 10 ml, EDTA tube 10 ml, SST tube 5 ml). Total blood drawing will be up to 55 ml in phase 1 patients and up to 82.5 ml in phase 2 patients. Serologic and additional immune assays will be conducted on blood drawn at these time points to assess for SARS-CoV-2 specific immune responses (see below).

ELIGIBILITY:
Inclusion criteria:

* Hospitalized patient (PUI or APS) and tested for SARS-CoV-2 by NP PCR swab
* At least one negative SARS-CoV-2 NP PCR swab within 2 wks of hospitalization
* Adult >/= 18 yrs old
* Patient or LAR provides informed consent
* Patient or LAR agree to follow-up procedures in informed consent form

Exclusion criteria:

* Prior reaction to blood drawing considered significant safety issue by study investigator
* Other factor considered significant safety issue by study investigator
* At least one positive SARS-CoV-2 NP PCR swab within 2 wks of hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients who have had pharyngeal testing negative for the presence of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 IgG | 120 days
  Qualitative seroconversion response rates (RR) in NP SARS-CoV-2 PCR swab negative PUI vs. swab negative APS patients will be compared as the primary outcome measurement.

SECONDARY OUTCOMES:
host immune response | 120 Days
  mRNA gene expression by RNAseq from whole blood collected into PAXGene RNA tubes
pathogen protein expression | 120 days
  identification of a signature of differentially expressed host genes or antigen/epitope specific antibody or cellular responses.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Freilich, MD, Principal Investigator — Bassett Medical Center
Locations (1):
- Bassett Medical Center, Cooperstown, New York, United States